CLINICAL TRIAL: NCT03851367
Title: Sling Suspension Versus Gym Balls in the Treatment of Juvenile Spinal Osteochondrosis in Adolescent Girls
Brief Title: Sling Suspension Versus Gym Balls in the Treatment of Juvenile Spinal Osteochondrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian Sports University (Other)
Collaborators: Lithuanian University of Health Sciences (Other); University of Brighton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LithuanianSportsU
Record Dates: First submitted 2019-02-20; First posted 2019-02-22 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Juvenile Osteochondrosis of Spine
Keywords: back pain; suspension therapy; Gymball; standing posture; muscle endurance
MeSH Terms: conditions — Scheuermann Disease; Back Pain

STUDY DESIGN:
Intervention Model Description: Subjects were recruited from an inpatient rehabilitation department, specializing in the treatment of children and adolescents with degenerative disorders. The research population consisted of 40 adolescents-girls, who were diagnosed with juvenile osteochondrosis (according to the International classification of Diseases - ICD M 42.0). All subjects were randomly divided into two groups: Sling Suspension Therapy, and Gymball therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sling suspension therapy (Experimental): 3-week duration of exercises using red cord and consisting of 15 sessions for 30 minutes each.
  Interventions: Procedure: Sling suspension using red cord
- Swiss ball therapy (Active Comparator): 3-week duration exercise for trunk muscles strengthening and posture improvement consisting of 15 sessions for 30 minutes each.
  Interventions: Procedure: Gym ball exercises

INTERVENTIONS:
Procedure: Sling suspension using red cord — 3 weeks duration, 15 sessions, and 30 minutes a day for five consecutive days a week. Back pain, endurance of trunk muscles (flexors, extensors and side flexors), and standing posture were evaluated pre and post interventions.
  Other Names: SST
  Arms: Sling suspension therapy
Procedure: Gym ball exercises — 3 weeks duration, 15 sessions, and 30 minutes a day for five consecutive days a week. Back pain, endurance of trunk muscles (flexors, extensors and side flexors), and standing posture were evaluated pre and post interventions.
  Other Names: GBT
  Arms: Swiss ball therapy

SUMMARY:
This study compares effect of swiss ball exercises with sling suspension exercises in the treatment of juvenile osteochondrosis in adolescent-girls

DETAILED DESCRIPTION:
One of the main tasks in the treatment of osteochondrosis related back pain is training trunk stabilizing muscles. This might be achieved by using a sling suspension exercise systems. Redcord is a trademark for Sling Exercise Therapy. Suspension exercise training has been shown to improves functional movement patterns more effectively than traditional exercise by creating a challenging and pain free environment for movement re-training. Another commonly used option in the treatment of juvenile osteochondrosis is Gymball, also known as Swissball core training programmes that are popular trends in physiotherapy and strength and conditioning programs. Benefits of Gymball core training exercises that facilitate spinal stability and balance have often been emphasized by researchers in development of strength and endurance, flexibility, and neuromuscular control as a cost effective and enjoyable way to treat and prevent back pain. Both exercises modes are used in treatment of back pain and muscle training in young people with juvenile osteochondrosis, what is why this study aims to compare Sling Suspension therapy with Gymball exercise in this population.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis - juvenile osteochondrosis (according to the International classification of Diseases - ICD M 42 gender: female

Exclusion Criteria:

* any other medical diagnosis

Ages: 14 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — only adolescents girls
Enrollment: 40 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Back pain | baseline
  was evaluated using the Visual Analogue Pain Scale (VAS). Participants were asked to report "current" pain intensity. A higher score indicates greater pain intensity: no pain (0-4 mm), mild pain (5-44 mm), moderate pain (45-74 mm), and severe pain (75- 100 mm).
Endurance of the trunk muscles | baseline
  was tested according those suggested by S. McGill (2007) and endurance duration was recorder in seconds. The back extensors ; The trunk flexors ; The lateral musculature
Weight | baseline
  Body weight was measured in kilograms with an accuracy of 100 g
Height | baseline
  Body height was measured in meters with an accuracy of 5 mm
Posture evaluation | baseline
  Standing posture was evaluated by a commonly used clinical assessment technique - visual assessment. In an attempt to minimize data collection error, one experienced examiner evaluated all the study participants' posture. The examiner was blind to the scope of the study and to the group that the subjects belonged to.

SECONDARY OUTCOMES:
Change in Back pain | 3 weeks
  was evaluated using the Visual Analogue Pain Scale (VAS). Participants were asked to report "current" pain intensity. A higher score indicates greater pain intensity: no pain (0-4 mm), mild pain (5-44 mm), moderate pain (45-74 mm), and severe pain (75- 100 mm).
Change in Endurance of the trunk muscles | 3 weeks
  was tested according those suggested by S. McGill (2007) and endurance duration was recorder in seconds. The back extensors ; The trunk flexors ; The lateral musculature
Improvement in Posture evaluation | 3 weeks
  Standing posture was evaluated by a commonly used clinical assessment technique - visual assessment. In an attempt to minimize data collection error, one experienced examiner evaluated all the study participants' posture. The examiner was blind to the scope of the study and to the group that the subjects belonged to.

CONTACTS AND LOCATIONS:
Locations (1):
- Vilma Dudoniene, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: Undecided
There is a plan to share IPD with other researchers